CLINICAL TRIAL: NCT01859702
Title: Pharmacokinetic Evaluation of Moxifloxacin in Vigadexa® in Aqueous Humor Samples Following Preoperative Antibiotic/Steroid Dosing in Cataract Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RDG-11-235
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-06

CONDITIONS: Cataract
Keywords: Aqueous Humor; Moxifloxacin; Vigadexa
MeSH Terms: conditions — Cataract | interventions — Moxifloxacin; Dexamethasone; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VIGADEXA (Experimental): Moxifloxacin 0.5%/Dexamethasone 0.1% ophthalmic solution, 1 drop instilled in the study eye 2 days before surgery, followed by 1 drop instilled 4 times a day the day before surgery. On the day of surgery, 1 drop was instilled 60 minutes prior to the procedure.
  Interventions: Drug: Moxifloxacin 0.5%/Dexamethasone 0.1% ophthalmic solution

INTERVENTIONS:
Drug: Moxifloxacin 0.5%/Dexamethasone 0.1% ophthalmic solution
  Other Names: Vigadexa®

SUMMARY:
The purpose of this study was to determine the moxifloxacin aqueous penetration when dosing with a combination drug Vigadexa preoperatively in cataract patients.

ELIGIBILITY:
Inclusion Criteria:

* Requires cataract surgery;
* Acceptable health status (medical history, physical, laboratory and ophthalmologic exams);
* Able to follow instructions and willing to attend all study visits;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any known or suspected allergies/hypersensitivity to any of the investigational test product components;
* History of invasive intraocular surgery in the eye to be operated, within 4 months before enrollment;
* Use of medications, as specified in protocol;
* Severe dry eye syndrome;
* Use of contact lenses two days before surgery until the last visit;
* External eye disease, infection or inflammation of the eyes or eyelids;
* Excessive bleeding tendency;
* No vision in the eye not included in the study;
* Pregnant or breastfeeding;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abayomi Ogundele, PharmD, Study Director — Alcon Research; Mauro Silveira de Queiroz Campos, MD, Principal Investigator — Federal University of São Paulo, Ophthalmology Service

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one study center in Brazil.
Pre-assignment Details: This reporting group includes all enrolled subjects.
Period: Overall Study
Arm/Group | VIGADEXA
Started | 36
Completed | 31
Not Completed | 5
Not completed — Protocol deviation | 3
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: This reporting group includes all enrolled subjects who received all doses of the test product.
Arm/Group | VIGADEXA
Number analyzed (Participants) | 35
Age Continuous [Mean (Standard Deviation); unit: years] | 71.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean Aqueous Humor Concentration of Moxifloxacin
Description: A 0.150 milliliter sample of the aqueous humor was obtained during cataract surgery. The concentration of moxifloxacin was measured by a validated procedure using high performance liquid-spectrometry.
Time Frame: Day 3 (operative day)
Population: Per protocol: All subjects who met inclusion/exclusion criteria, received all doses of the test product, and underwent cataract surgery with aqueous humor sampling.
Measure: Mean (95% Confidence Interval); unit: nanograms per milliliter
Arm/Group | VIGADEXA
Number analyzed (Participants) | 31
nanograms per milliliter | 1110.6 [857.5 to 1363.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. An adverse event was defined as any untoward medical occurrence, or deterioration of a pre-existing medical condition, that occurred during or after test product administration.
Description: Adverse events were obtained as solicited comments from the study subjects and as observations by the study Investigator as outlined in the study protocol.
Arm/Group | VIGADEXA
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 2/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VIGADEXA (N=36)
Hypertensive Crisis (Cardiac disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.